CLINICAL TRIAL: NCT04190069
Title: Effects of Behavioral Interventions on Weight Loss and Weight Maintenance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB recommended change to registry study or quality improvement project status
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Rometo, Clinical Director for UPMC Center for Obesity Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY19100189
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Behavior
Keywords: weight loss, weight maintenance
MeSH Terms: conditions — Behavior; Weight Loss | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIFAST only (No Intervention): Control group will consist of participants that have not undergone behavioral modifications with the Prescription for Wellness Program. These are participants that only go through the OPTIFAST Program.
- UPMC PFW followed by OPTIFAST (Experimental): The intervention group will consist of participants that have undergone behavioral modifications with the Prescription for Wellness Program. These are participants who undergo the Prescription for Wellness Program prior to the OPTIFAST Program.
  Interventions: Behavioral: Behavioral interventions/modifications

INTERVENTIONS:
Behavioral: Behavioral interventions/modifications — UPMC Prescription for Wellness is an innovative physician/provider prescribed coaching and feedback program that improves patient engagement and outcomes in healthy behaviors; self-care of chronic disease and condition management; and shared decision-making. The resources available through this program are offered via a telephonic health coach, online or through a digital intervention based on the participant's convenience.
  Arms: UPMC PFW followed by OPTIFAST

SUMMARY:
The objective of the study is to examine the extent to which diet/lifestyle change programs with a multidisciplinary team (consisting of a dietician, physician and behaviorist/health coach) that develop healthy behaviors before creating a calorie deficit for weight loss will result in greater weight loss and a longer duration of weight maintenance. It intends to compare the extent of weight loss and weight maintenance in participants who will undergo calorie restriction without prior behavioral interventions to participants that will undergo behavioral interventions prior to starting calorie restriction.

DETAILED DESCRIPTION:
OPTIFAST is a medically supervised weight loss and weight management program that involves a complete meal replacement followed by a gradual introduction of foods after dietary education. The resources offered through this program are through a physician, registered dietitian and behaviorist, including a psychologist.

UPMC Prescription for Wellness is an innovative physician/provider prescribed coaching and feedback program that improves patient engagement and outcomes in healthy behaviors; self-care of chronic disease and condition management; and shared decision-making. The resources available through this program are offered via a telephonic health coach, online or through a digital intervention based on the participant's convenience.

The objective of the study is to examine the extent to which diet/lifestyle change programs with a multidisciplinary team (consisting of a dietician, physician and behaviorist/health coach) that develop healthy behaviors before creating a calorie deficit for weight loss will result in greater weight loss and a longer duration of weight maintenance. It intends to compare the extent of weight loss and weight maintenance in participants who will undergo calorie restriction without prior behavioral interventions to participants that will undergo behavioral interventions prior to starting calorie restriction.

Behavioral interventions will first be provided by UPMC Prescription for Wellness prior to starting OPTIFAST. Calorie restriction will be during the OPTIFAST Program. The participants will be actively recruited by the study team at the Center for Diabetes and Metabolism (CDE) at the Falk Clinic in Oakland, Pittsburgh.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 yrs or older
2. BMI >40 kg/m2
3. BMI between 35-40 kg/m2 with obesity-related co-morbidities including type 2 diabetes mellitus, hypertension, dyslipidemia. Type 2 Diabetes Mellitus defined by A1c >6.4% with or without oral hypoglycemic agents and with or without insulin therapy. Hypertension defined by blood pressure >140/80 mm of hg with or without antihypertensive therapy. Dyslipidemia defined as fasting lipid profile with one or more of the following abnormalities: serum cholesterol levels >200 mg/dl, serum triglyceride levels >150 mg/dl, HDL levels <50 mg/dl, LDL levels >100 mg/dl with or without therapy.

Exclusion Criteria:

1. Binge eating disorder (Bulemia, Anorexia nervosa)
2. Congestive heart failure NYHA Class >3
3. >Stage 3 chronic kidney disease
4. Cardiovascular disease (non-fatal MI, non-fatal stroke, peripheral vascular disease) within the past 6 months of screening
5. Planned coronary artery, carotid artery or peripheral artery revascularization
6. Weight loss surgery (gastric bypass, sleeve gastrectomy, total/subtotal gastrectomy) within the past 2 yrs.
7. Pregnant and lactating females
8. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight at 6 months | 6 months
  The degree of weight loss in those who undergo behavioral modifications prior to starting calorie restriction compared to those who do not undergo behavioral modifications prior to starting calorie restriction.
Change from 6 months in body weight at 18 months | 6 months vs 18 months
  The duration of weight maintenance in those who undergo behavioral modifications prior to starting calorie restriction compared to those who do not undergo behavioral modifications prior to starting calorie restriction.

SECONDARY OUTCOMES:
Change from baseline in blood pressure at 18 months | 18 months
  change in blood pressure over time in participants who undergo behavioral interventions compared to those who do not.
Change from baseline in A1c at 18 months | 18 months
  change in A1c over time in participants who undergo behavioral interventions compared to those who do not.
Change from baseline in lipid profile at 18 months | 18 months
  change in lipid profile overtime in participants who undergo behavioral interventions compared to those who do not.
Change from baseline in medication burden (number of medications) at 18 months | 18 months
  Change in medication burden (number of medications) pertaining to type 2 DM and hypertension over time
Change from baseline in medication burden (dose of medications) at 18 months | 18 months
  Change in medication burden (dose of medications) pertaining to type 2 DM and hypertension over time

CONTACTS AND LOCATIONS:
Overall Officials: David Rometo, M.D, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No